CLINICAL TRIAL: NCT03608449
Title: Doing More With Less": Optimizing Psychotherapeutic Services in the Mental Health System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SHA-005-18
Record Dates: First submitted 2018-07-08; First posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Anxiety Disorder; Affective Disorders; Personality Disorders
MeSH Terms: conditions — Anxiety Disorders; Mood Disorders; Personality Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Parallel, randomized by order, open study, assignment (matching/rematching) supported by monitoring data.
Masking Description: not relevant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Active Comparator): after monitoring treatment outcomes for 4 weeks, treatment plan or psychotherpist will be changed according to scoring by the director of department.
  Interventions: Other: questionnaires
- control group (Placebo Comparator): treatment as usual. treatment counitunes as usual without depending on monitoring treatment outcomes.
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires — questionnaire about mental health status during psychotherapy

SUMMARY:
Psychotherapy is one of the cornerstones of mental health services. It is provided by psychiatrist, psychologists and psychiatric social worker in both hospital and out-patient services, and is assumed to require massive manpower and training inputs.

Internationally, the clinical outcomes of routine mental health services are rarely recorded or reported. However, a rough estimation is that half (40-60%) of all psychotherapies have a favorable clinical outcome. Recently (Clark et al, 2017), the English Improving Access to Psychological Therapies (IAPT) Program, which delivers psychotherapies to more than 537 000 patients in the UK each year, indicated that 44% of the patients recovered, and 62%- improved. Consistent with a causal model, most organizational factors also predicted between-year changes in outcome, together accounting for 33% of variance in reliable improvement and 22% for reliable recovery.

The proposed study aims at dramatically improving the yield of psychotherapies in the Mental Health Services by combining monitoring and patient-therapist matching strategies. The first will be achieved by implementing Routine Outcome Monitoring (ROM), and the second- by applying a patient-therapist match-re-match procedure during psychotherapy

DETAILED DESCRIPTION:
Routine Outcome Monitoring Routine Outcome Monitoring (ROM) enables systematic assessment of treatment outcomes at regular intervals for monitoring the progress of patients during treatment. ROM was originally developed for clinical studies, thus providing quality feedback for research and clinical purposes. There is accumulated evidence that ROM has positive effects for supporting care, for research and for management.

As of the beginning of the previous decade, ROM projects have developed and integrated into national health systems (e.g. Australia and New Zealand, England, etc.) and in various research groups around the world (e.g. Holland, Italy, USA, Canada, (Ruggeri, 2002; Burgess et al., 2012; Mellor-Clarket al., 2006) .In recent years, computer software has been widely used to collect, analyze and manage information in a secure, efficient and accessible manner, providing ongoing feedback to caregivers (Barkham et al., 2001; Barkham & Mellor-Clark, 2003; Margison et al., 2000).

Routine outcome monitoring can enable achieving several goals that directly contribute to treatment (De Beurs et al., 2011). It provides quality feedback to clinicians and patients in real time about the progress of the treatment and the early identification of various problems such as negative response to therapy. This increases the positive response to the treatment, balances the therapist's biases in an optimistic or pessimistic direction, supports decisions in treatment and improves the cooperation between the therapist and the patient. Hence, patients' involvement in the therapeutic process, their commitment to it, and their satisfaction (Whipple & Lambert, 2011), Lambert, 2010 (Priebe et al., 2002) also improve. A group of studies has shown that frequent monitoring of the evaluation of the therapeutic relationship during psychotherapy enables better real-time identification of therapeutic ruptures that can be corrected (Muran et al. 2009; Safran et al., 2011). In psychiatric work with more severe patients, it was demonstrated that there was a correlation between ROM and a significant reduction in the number and duration of hospitalizations, a finding that has a significant economic significance (Slade et al., 2006). In a meta-analysis review published in 2009 (12 studies, 2001-2006) a significant short-term symptomatic improvement and some long-term improvements was shown in monitored therapies. In another review (Shimokawa et al., 2010), a weekly measure of personal well-being measures had a significant positive impact on the quality, duration and outcome of treatment, especially in patients prone to dropout. Despite initial objections among teams to introduce quantitative measurements into their work, various attempts have shown that after assimilation, staff satisfaction from the systems is great and serves as a complement to individual work and staff meetings (de Beurs et al., 2011).

The collection of the broad information in the ROM is also used for managerial purposes (Trauer, 2010). For example, the accumulated information can be used for ongoing epidemiological research of treatments as they actually occur in a heterogeneous clinical environment and may maximize resources utilization (Coombs et al., 2011). The information produced (on the organizational, local, regional or national levels) is more likely to have higher predictive validity than information extracted from incidental questioning patients for improvement. Effective evaluations of various treatment approaches have also been made, and it is important to consider that treatments are indeed effective in the particular clinical setting they are provided, and not only in controlled studies under very different conditions (Stiles et al., 2008). Applying ROM appears to be more effective when integrated in a formalized and structured manner (Krägeloh, 2015). In such terms, it may be a powerful managerial tool, balancing between the patient's expectations and needs and the mental health care capacity. It is thus surprising, as recently noted by Jensen-Doss (2018), that ROM rarely used in practice, even though it is viewed favorably.

Despite current enthusiasm, advances in implementation, and the growing belief among some proponents and policymakers that ROM represents a major revolution in the practice of psychotherapy, other research has suggested that the focus on measurement and monitoring is in danger of missing the point (Miller et al., 2015). Research from the field of expertise and expert performance provides guidance for realizing the full potential of ROM. One crucial element in optimizing the effect of the ROM is that the decisions derived from continuously collecting the outcome measures will be taken with the patient (and not just shared with him/her). As shown by Clarke et al. (2015), more active involvement in decision-making than the patient stated as desired was associated with higher satisfaction. A clinical orientation towards empowering, rather than shared, decision-making may maximize satisfaction and optimize the effect ROM may have on clinical practice.

Implementation of novel strategies in the field of psychiatry may result in substantial cost reduction (van Londen, 2016) Patient-therapist matching in psychotherapy Research on fitting treatment procedures to the unique needs and proclivities of patients is limited. Traditional research on efficacy of psychotherapy focuses on the role of interventions and theoretical brands, minimizing factors that cannot be randomly assigned. This line of research has not realized its initial and desired promise, perhaps because it fails to incorporate into the study of psychotherapy important and effective treatment variations that are associated with therapist and non-diagnostic patient factors (Beutler, 2015).

The possibility to match patient to therapist by pre-treatment data did not succeed. Many factors were found to contribute to good outcome in psychotherapies. These include patient's factors (e.g.- high levels of motivation and involvement with positive, but realistic attitude), therapist's factors (e.g.- training and supervision) and relational factors (strength of therapeutic alliance is a leading factor; other factors are of moderate- to poor-correlation to outcome) (Cooper, 2008).

While it is accepted that pre-treatment patient-therapist match will not do, the possibility to re-match patient-therapist dyads in case of unsuccessful therapies clinically sounds. Surprisingly, to our best knowledge, this possibility was never examined. Thus, while the ROM clearly indicates whether the trajectory of a given psychotherapy is favorable, it is not examined for initiating patient-therapist re-matching in therapies with poor outcome. This can be attributed to the personal and protected nature of the psychotherapy, generally perceived as indifferent to external observation.

RESEARCH ASSUMPTIONS Co-implementation of patient- and therapist-based routine monitoring tools with matching/re-matching strategies will promote therapy outcome in 25% and will not reduce total patients' satisfaction.

As measured in cost-effectiveness values, our secondary assumption is that co-implementation of monitoring-&-managing systems will reduce 28% of mental health costs in the unit examined.

STUDY DESIGN The study (see Figure 1 attached at the end of the proposal) will span over 21 months, of which 14 months will be dedicated for assessing the effect of monitoring-&-matching system in one out-patient intensive mental health facility.

The study will be performed in the Day Care Department (DCD) of the Shalvata Mental Health Center (SMHC). This unit treats patients who suffer from psychiatric disorders but do not require full hospitalization. The DCD is part of the SMHC out-patient network, and admits patients directly from the community (half-way in). The department has a diverse team (30 professionals) of psychiatrists, psychologists, social workers, occupational therapists, expressive therapists and nursing staff, and receives about 10-15 patients each month. The DCD is ideal for testing new therapeutic strategies in the field of psychiatry: it supplies intensive care (thus enabling frequent monitoring of the patient's condition), it operates in large volumes (i.e., can quickly examine proposals for implementing treatment systems), it is backed by sophisticated information systems (Chameleon; an integrated electronic medical record system) and as it is situated "in-between" the hospitalizing and ambulatory systems (it covers both of them).

The proposed study in a pilot study, thus focusing on a relatively small number of participants. Altogether, one hundred patients will be enrolled in the study, randomized-by-order to either the monitored-&-matched ("re-matched") group, or the treated-as-usual (TAU) group. Enrolled patients of the two groups will be followed for their entire day-care period, or to a period of 3 months (the shorter of the two). Follow up will include in both re-matched and TAU groups formalized (SCID) and an array of self-reported questionnaires (see below). Patients and therapists of the both group will routinely complete ROM questionnaires, as well as mid- and end-term questionnaires evaluating their condition and satisfaction; only patients of the re-matched group will be matched/re-matched (see below).

ELIGIBILITY:
Inclusion Criteria:

1. All enrolled patients must have a mobile phone capable of hosting the ROM-on-mobile system.
2. patients with anxiety/ affective (depressive and bi-polar)/ personality disorders

Exclusion Criteria:

1. Patients exceeding 65 years at their date of admission,
2. Patients with impaired Hebrew fluency (difficulties in either reading or writing),
3. Evidence of organic brain syndrome or mental retardation,
4. Patients with psychotic disorders (e.g. - schizophrenia, delusional disorders)
5. Evidence of probable need for hospitalization,
6. Patients admitted only for diagnostic purposes,
7. Patients unwilling to be enrolled in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
OQ-45 (outcome measure) | up to 14 months
  is the most commonly-used outcome measure in psychotherapy. It provides both a measure of weekly change on which the feedback to therapists and patients was based and the criterion measure for classification of a patient into an outcome group on a scale of 0 ("never") to 4 ("always")
SEQ (session outcome) | up to 14 months
  The SEQ-4 validates the WAI-6, and allows the better identification of sessions in which ruptures and repairs occurred. The questionnaire includes 20 bipolar statements ranges on a 7 degrees Likert scale (e.g.:, 1 "sad" to 7 "happy"). the statements refers to 2 dimensions: the dimension of the meeting itself ("the current meeting was ...") and the dimension of feeling ("I feel now ...").
WAI (working alliance) | up to 14 months
  To measure alliance at the end of each session, we will use the patient-version of the Session Alliance Inventory. The SAI is a 6-item short-short version of the Working Alliance Inventory. the questionnaire includes 6 items on a scale of 1 ("does not describe how I feel") to 7("exactly describes how I feel").
HSCL-11 (symptoms) | up to 14 months
  The HSCL-11 will be filled by the patient at the beginning of study and thereafter- every two weeks. it includes 11 items on a scale of 1 ("not at all") to 4("a lot").

SECONDARY OUTCOMES:
PWB (psychological well-being) | up to 14 months
  The PWB , filled by the patient at the beginning of study and thereafter- every two weeks, in a commonly used questionnaire assessing psychological well-being with acceptable psychometric properties and convergence with prior indexes of well-being. it includes 54 items ranked on a scale of 1("don't agree") to 6 ("very much agree").
Satisfaction from therapy (CSQ) | up to 14 months
  . The CSQ is a standardized measure with strong psychometric properties that could be used to assess general satisfaction across varied health and human services.

CONTACTS AND LOCATIONS:
Overall Officials: Shlomo Mendalovitch, Dr, Principal Investigator — Shalvata mental health hospital

IPD SHARING:
Plan to Share IPD: No
no plan